CLINICAL TRIAL: NCT01408485
Title: Clinical Evaluation of Therapy™ Cool Flex™ Irrigated Ablation System for the Treatment of Typical Atrial Flutter
Brief Title: Therapy™ Cool Flex™ Irrigated Ablation System for Typical Atrial Flutter
Acronym: FLEXION-AFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90067869
Record Dates: First submitted 2011-07-22; First posted 2011-08-03 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Typical Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Radio-frequency cardiac ablation for treatment of isthmus-dependant atrial flutter using the Therapy™ Cool Flex™ Irrigated Ablation System
  Interventions: Device: Therapy™ Cool Flex™ Irrigated Ablation System

INTERVENTIONS:
Device: Therapy™ Cool Flex™ Irrigated Ablation System — The investigational components of the Therapy™ Cool Flex™ Irrigated Ablation System consist of:
  * Therapy™ Cool Flex™ 4mm Irrigated Ablation Catheter
  * IBI 1500T9 V1.43 RF Generator

SUMMARY:
To demonstrate that ablation with the Therapy™ Cool Flex™ Irrigated Ablation System is effective in the treatment of typical atrial flutter (cavo-tricuspid dependent) and that its use does not result in an unacceptable risk of intra-procedural, serious cardiac adverse events.

DETAILED DESCRIPTION:
This will be a prospective, multi-center and non-randomized study. All treated patients will receive ablation therapy for typical atrial flutter using the TherapyTM Cool FlexTM Irrigated Ablation System. Historical data from combined published (PMA P060019 Cool Path) and reported (IDE G090109 Cool Path Duo) Atrial Flutter studies will be used to determine performance goals for study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* A signed written Informed Consent
* Presence of typical atrial flutter (cavo-tricuspid isthmus dependent)
* If subjects are receiving anti-arrhythmic drug therapy (Class I or Class III AAD) for an arrhythmia other than typical atrial flutter, then the subject needs to be controlled on their medication for at least 3 months. If the subject had typical atrial flutter before starting the AAD(s) (Class I or Class III) and then subsequently had another arrhythmia (i.e. atrial fibrillation), then the 3 month AAD criteria will not apply
* One documented occurrence of the study arrhythmia documented by ECG, Holter, telemetry strip, or transtelephonic monitor within the past 6 months
* In good physical health
* 18 years of age or older
* Agree to comply with follow-up visits and evaluation

Exclusion Criteria:

* Prior typical atrial flutter ablation treatment
* Pregnancy
* Atypical flutter or scar flutter (non isthmus dependent)
* Significant coronary heart disease or heart failure; that is unstable angina pectoris and/or uncontrolled congestive heart failure (NYHA Class III or IV) at the time of enrollment
* A recent myocardial infarction within 3 months of the intended procedure date
* Permanent coronary sinus pacing lead
* Clinically significant Tricuspid valvular disease requiring surgery and/or a prosthetic tricuspid heart valve
* Evidence of intra-cardiac thrombus or a history of clotting disorders
* Participation in another investigational study
* Cardiac surgery within 1 month prior to the intended procedure date
* Allergy or contraindication to Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Weiss, MD, Principal Investigator — Ohio State University
Locations (24):
- United States (22):
  - St. Joseph's Hospital-Heart Rhythm Specialists, PC, Phoenix, Arizona
  - Summit - Cardiovascular Consultants Med Group, Inc., Oakland, California
  - Huntington Memorial / Foothill Cardiology, Pasadena, California
  - Regional Cardiology Associates, Sacramento, California
  - Community Memorial Hospital, Ventura, California
  - Adventist Health / Florida Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Joseph's Hospital, Atlanta, Georgia
  - Washington Hospital Center, Georgetown, Maryland
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Jersey Shore Universty Medical Center, Neptune City, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Cleveland Clinic / Cardiovascular Associates of Cleveland, Mayfield Heights, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Sacred Heart Med Center, Springfield, Oregon
  - Guthrie-Robert Packer Hospital, Sayre, Pennsylvania
  - Clinical Tex Research, LLC/DBA PharmaTex Research, Amarillo, Texas
  - Heart Hospital of Austin, Austin, Texas
  - Methodist Hospital Research Institute, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
- Canada (2):
  - VCAT / Royal Jubilee, Victoria, British Columbia
  - Institut de Cardiologie de Quebec (Hopital Laval), Québec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 200
Completed | 179
Not Completed | 21
Not completed — Withdrawal by Subject | 21

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.28 (10.18)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 89
  >=65 years | 111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 158
Region of Enrollment [Number; unit: participants]
  United States | 182
  Canada | 18

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety: Incidence of Composite, Serious Adverse Events Within 7 Days Post-Procedure
Description: Primary safety is defined as the incidence of composite, serious adverse events within 7 days post-procedure, regardless of whether a determination can be made regarding device relatedness.
Time Frame: 7 days
Population: 200 subjects who met Inc/Excl criteria were enrolled. 21 subjects were withdrawn prior to the use of the investigational device, thus, 179 were treated. 5 subjects had composite adverse events that were serious and occurred within 7 days of the ablation procedure. These events are part of the primary safety endpoint analysis per protocol.
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 179
participants | 5

2. Primary Outcome: Primary Efficacy
Description: Primary efficacy or acute success is defined as achievement of bi-directional block in the cavo-tricuspid isthmus and non-inducibility of typical atrial flutter at least 30 minutes following the last RF ablation with the investigational system.
Time Frame: 30 minutes
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 179
participants | 177

3. Secondary Outcome: Secondary Efficacy
Description: Secondary efficacy or chronic success is defined as freedom from recurrence of typical atrial flutter 3 mos. post ablation. Flutter recurrence will be documented on an ECG. Repeat ablations, new antiarrhythmia medications or increase in the existing anti-arrhythmic medications during the 3 mos. post ablation are considered chronic failures.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 175
participants | 150

ADVERSE EVENTS:
Description: 200 subjects who met Inc/Excl criteria were enrolled. 21 subjects were withdrawn prior to the use of the investigational device, thus, 179 were treated. 5 subjects had composite adverse events that were serious and occurred within 7 days of the ablation procedure. These events are part of the primary safety endpoint analysis per protocol.
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 5/179
Other Adverse Events (participants affected / at risk) | 9/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=179)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Arrythmia (Cardiac disorders) | 1 (1)
Other (General disorders) | 1 (1) — Death event
Stroke/Cerebrovascular Accident (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=179)
Palpitations (Cardiac disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other